CLINICAL TRIAL: NCT01466920
Title: Why Are so Many Patients Dissatisfied With Knee Replacement Surgery? Exploring Variations of the Patient Experience
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H11-02117
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Total Knee Arthroplasty
Keywords: Total knee arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The goal of this research is to fill the knowledge gap relating to why up to 20 percent of total knee arthroplasty (TKA) patients are dissatisfied with their clinical outcomes and to answer the research question: What are the drivers of variation in the patient experience with primary (ie. not revision) TKA?

DETAILED DESCRIPTION:
Purpose: Among patients with a diagnosis of osteoarthritis and who are undergoing total knee arthroplasty:

1. To identify variations in the patient experience with primary knee replacement surgery by measuring clinical outcomes, health status, and patient satisfaction; and
2. To explore the factors contributing to good/poor clinical and patient outcomes, such as surgical factors, health system factors, socioeconomic demographic factors and psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 and older
* Primary or secondary diagnosis of osteoarthritis or inflammatory arthritis
* Scheduled to undergo primary TKA
* Living in British Columbia
* Capable of providing informed consent

Exclusion Criteria:

* Not having been diagnosed with osteoarthritis
* Inability to complete the study questionnaires
* Adults undergoing arthroplasty revision surgery
* Adults undergoing bilateral knee replacements
* Adults undergoing unicompartmental knee replacements
* Adults whose knee replacement is due to post-traumatic deformity Contacts and Locations

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stirling Bryan, PhD, Principal Investigator — School of Population and Public Health, University of British Columbia; Jennifer Davis, PhD, Study Director — University of British Columbia; Alison Dormuth, Study Director — BC Ministry of Health Services; Denise Dunton, MN, Study Director — Interior Health Authority; Vivian Giglio, Study Director — Fraser Health Authority; Laurie Goldsmith, MSc, PhD, Study Director — Simon Fraser University; Val MacDonald, MSN, Study Director — Fraser Health Authority; Patrick McAllister, MD, Study Director — Vancouver Island Health Authority; Rick Sawatzky, PhD, RN, Study Director — Trinity Western University
Locations (7):
- Canada (7):
  - Burnaby Hospital, Burnaby, British Columbia
  - Kelowna General Hospital, Kelowna, British Columbia
  - University Hospital of Northern British Columbia, Prince George, British Columbia
  - Richmond Hospital, Richmond, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia
  - VIHA Joint Replacement Clinic, Victoria, British Columbia